CLINICAL TRIAL: NCT04848909
Title: Post-Prostatectomy Linac-Based Ultrahypofractionated Radiotherapy for Patients With Localized Prostate Cancer: A Treatment Feasibility and Outcomes Multicenter Study
Brief Title: Stereotactic Body Radiotherapy (SBRT) Post Prostatectomy
Acronym: PLUTO-MPC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Royal Victoria Regional Health Centre (Unknown); Princess Margaret Hospital, Canada (Other); Credit Valley Hospital (Other)
Responsible Party: Principal Investigator, Chia-Lin (Eric) Tseng, Principal Investigator, Assistant Professor, Dept of Radiation Oncology Sunnybrook Odette Cancer Centre, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3596
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: SBRT; Ultrahypofractionated Radiotherapy; Localized Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: men diagnosed with prostate cancer post-prostatectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Men with prostate cancer post-prostatectomy (Experimental): Men with localized prostate cancer who are considered candidates for post-prostatectomy radiation.
  Interventions: Radiation: stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: stereotactic body radiotherapy (SBRT) — Stereotactic body or external-beam radiation therapy (SBRT) is a method of delivery of radiation in precision manner to the prostate bed in this study. The SBRT dose prescription will be 3000 cGy in 5 fractions to the prostate bed and 2500 cGy in 5 fractions to the pelvic nodes if elective nodal irradiation (ENI) is used, delivered every other business day.

SUMMARY:
This phase I study will assess the toxicity profile and efficacy of SBRT (Stereotactic body radiotherapy) in patients with localized prostate cancer who are considered candidates for post-prostatectomy radiation.

DETAILED DESCRIPTION:
Radical prostatectomy is a common treatment for localized prostate cancer, patients with a detectable and/or rising PSA after radical prostatectomy may be offered radiation. An increasing number of patients are being referred post-operatively for radiotherapy, which creates an added burden on radiotherapy departments. Therefore, a strategy that could potentially decrease the number of radiotherapy fractions, yet maintain its efficacy, would be highly desirable for patient convenience, cost saving, and resource utilization as long as the toxicity profile is acceptable. This study will be conducted to asses the toxicity and efficacy of Stereotactic body radiotherapy (SBRT) in post-prostatectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate status post radical prostatectomy
* Completed written informed consent
* Able and willing to complete EPIC, PORPUS, and EQ-5D questionnaires
* A detectable PSA ≤ 2.0 ng/ml
* Two consecutive rises in PSA and final PSA > 0.1 ng/ml OR three or more consecutive rises in PSA

Exclusion Criteria:

* Gross residual disease (per conventional imaging, i.e. CT and/or MRI)
* Histological or radiological node +ve (N1) or distant metastases (M1)
* Prior pelvic radiotherapy
* Contraindications to radical pelvic radiotherapy (e.g. connective tissue disease or inflammatory bowel disease)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Early Adverse Events/toxicities experience by Participants | 6.5 years
  Incidence of acute GU and GI toxicities, based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Late Adverse Events/toxicities experienced by Participants | 6.5 years
  Incidence of late GU and GI toxicities (≥6 months) using CTCAE v5.0
Quality of Life of participants using the Expanded Prostate Cancer Index Composite questionnaire | 6.5 years
  Acute and late GU and GI quality of life (QoL) using the Expanded Prostate Cancer Index Composite questionnaire which evaluates participant's function and bother after prostate cancer treatment. Each question is scored from 1-5, 1 being the better outcome and 5 being the worst outcome.
Biochemical disease-free survival | 6.5 years
  Biochemical disease-free survival (bDFS), defined as survival until first evidence of either biochemical progression (PSA of 0.4 ng/mL or greater) following postoperative radiotherapy, PSA of more than 2.0 ng/mL at any time after postoperative radiotherapy, clinical or radiological progression, initiation of non-protocol hormone therapy, or death from prostate cancer
Health Utilities using The Patient-Oriented Prostate Utility Scale | 6.5years
  Health utilities using The Patient-Oriented Prostate Utility Scale to measure health-related quality of life, whether it improves, deteriorates or stay the same. There are 10 questions, each questions has 5 possible answers, with 1 being the better outcome and 5 being the worst outcome.
Health Utilities using EuroQol- 5 Dimension Questionnaire | 6.5years
  Health utilities using the EuroQol- 5 Dimension Questionnaire determines 5 variables, each with 5 possible options, with the first being the best outcome and the last being the worst outcome. The 5 variables include:
  1. Mobility
  2. Self-care
  3. Usual Activities
  4. Pain/discomfort
  5. Anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Chia-Lin Tseng, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Onatrio, Canada

IPD SHARING:
Plan to Share IPD: No